CLINICAL TRIAL: NCT03870373
Title: Validate Pulse Oximeter Sensors in Neonates by Comparing Sensor Readings to Blood Samples During Cardiac Surgery
Brief Title: Performance of Pulse Oximeter Sensors in Neonates
Status: Completed | Type: Observational
Sponsor: Taiwan Aulisa Medical Devices Technologies, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 18-25904
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Test Subject: neonatal patients undergoing complex cardiac surgical procedures
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter — Aulisa's non-invasive pulse oximeter sensor is applied to a foot of the neonate; an adhesive patch secures the sensor to the neonate.

SUMMARY:
Validate pulse oximeter sensors in neonates by comparing sensor readings to blood samples during cardiac surgery.

DETAILED DESCRIPTION:
Researchers at the University of California, San Francisco have developed methods that permit them to test multiple pulse oximeter sensors on neonates simultaneously during cardiac surgery. During this type of surgery, the arterial oxygen saturation changes over a wide range, providing an ideal arena for the assessment of neonatal pulse oximeter sensors at many levels of oxygen saturation. Several arterial blood gas samples are typically obtained during these procedures. Saturation of each arterial blood sample is determined by direct oximetry in a hemoximeter and this measurement is compared to the reading displayed on the pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Neonates scheduled to undergo cardiac surgery where routine blood draws would be taken
* Consent signed by at least one legal guardian

Exclusion Criteria:

* Presence of any skin irritation or breakdown on the foot
* Foot impediments which would preclude proper placement of the sensor
* Clinical condition precluding the use of adhesive materials

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal patients undergoing complex cardiac surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Performance of Pulse Oximeter Sensor in Neonates | Data are collected anywhere from the beginning of surgery until the completion of the procedure
  Pulse Oximeters - Premarket Notifications Submissions [510(k)s] Guidance For Industry and Food and Drug Administration Staff (issued: March 4, 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Hung G Nguyen, MD, Principal Investigator — UCSF Medical Center at Mission Bay
Locations (1):
- UCSF Medical Center at Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided